CLINICAL TRIAL: NCT01513798
Title: Diet and Exercise in Type 2 Diabetes - a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Tommy Olsson, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2011-294-31M
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diet Therapy; Exercise Therapy; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Exercise under observation (Experimental): Modified paleolithic diet and exercise 3 sessions/week under observation
  Interventions: Behavioral: Modified paleolithic diet and exercise under observation
- General advice on exercise (Experimental): Modified paleolithic diet and general advice on exercise
  Interventions: Behavioral: Modified paleolithic diet and general advice on exercise

INTERVENTIONS:
Behavioral: Modified paleolithic diet and exercise under observation — Modified paleolithic diet and exercise 3 session/week under observation
  Arms: Exercise under observation
Behavioral: Modified paleolithic diet and general advice on exercise — Modified paleolithic diet and general advice on exercise
  Arms: General advice on exercise

SUMMARY:
The investigators investigate if combined progressive aerobic training and resistance training improve metabolic control and fat mass in patients with type 2 diabetes who are eating a modified paleolithic diet. The investigators randomize 40 participants to two groups: 1) Modified paleolithic diet and exercise under observation 3 sessions/week, 2) Modified paleolithic diet and general advice about exercise.

The investigators primary hypothesis is that in patients with type 2 diabetes decreases fat mass more with progressive exercise under observation and a modified paleolithic diet than with general advice about exercise and a modified paleolithic diet.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes less than 10 years
* BMI 27-35
* women only after menopause
* diabetes treatment with diet and/or metformin
* HbA1c between 45 and 94

Exclusion Criteria:

* nicotine use
* insulin
* betablockers
* estrogens orally
* blod pressure >160/100
* macroalbuminuria
* malignancy during the past 5 years
* alcoholism
* depression
* cardiovascular disease/stroke
* liver disease
* serious lung disease, GI disease or kidney disease
* more than 30 minutes/5 days a week of moderate exercise during the last 6 months
* resistance training during the past 6 months
* official weight loosing program during the past year
* obesity surgery
* night work
* MADRS-S (Montgomery Asberg Depression Rating Scale) >20 points
* AUDIT >14 points for women, >16 points for men
* not possible to obtain venous sampling

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Fat mass | Baseline - 12 weeks
  Measured with DEXA (dual energy x-ray absorptiometry)

SECONDARY OUTCOMES:
Peripheral insulin sensitivity | Baseline - 12 weeks
  Measured with euglycemic hyperinsulinemic clamp
Hepatic insulin sensitivity | Baseline - 12 weeks
  Measured with euglycemic hyperinsulinemic clamp
Liver fat | Baseline - 12 weeks
  Measured with 1H-MRS (proton magnetic resonance spectroscopy)
Cortisol turnover | Baseline - 12 weeks
Appetite regulation | Baseline - 12 weeks
  GLP-1 (glucagon-like peptide 1), peptide YY
Dopamine 2-receptors in striatum | Baseline - 12 weeks
  PET
Executive ability and memory | Baseline - 12 weeks
  fMRI (functional magnetic resonance imaging)
Experience of training | Baseline - 12 weeks
  SCI ESES (Spinal Cord Injury Exercise Self-Efficacy Scale, ABC (Activities-specific Balance Confidence scale), PRETIE-Q (Preference for and Tolerance of the Intensity of Exercise Questionnaire)
Validity of energy intake and protein intake | Baseline - 6 weeks - 12 weeks
  Actiheart®, food diary, weight, nitrogen excretion
Oxygen Uptake | Baseline - 12 weeks
  Cardiopulmonary exercise testing
Anaerobic Threshold | Baseline - 12 weeks
  Cardiopulmonary exercise testing
Substrate utilization during submaximal exercise | Baseline - 12 weeks
  Measured with indirect calorimetry during ergometer cycling

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Olsson, Professor, Principal Investigator — Department of Public Health and Clinical Medicine, Umeå University
Locations (1):
- Department of Public Health and Clinical Medicine, Medicine, Umeå, Sweden

REFERENCES:
- [Derived] Otten J, Andersson J, Stahl J, Stomby A, Saleh A, Waling M, Ryberg M, Hauksson J, Svensson M, Johansson B, Olsson T. Exercise Training Adds Cardiometabolic Benefits of a Paleolithic Diet in Type 2 Diabetes Mellitus. J Am Heart Assoc. 2019 Jan 22;8(2):e010634. doi: 10.1161/JAHA.118.010634. PMID 30652528
- [Derived] Otten J, Stomby A, Waling M, Isaksson A, Soderstrom I, Ryberg M, Svensson M, Hauksson J, Olsson T. A heterogeneous response of liver and skeletal muscle fat to the combination of a Paleolithic diet and exercise in obese individuals with type 2 diabetes: a randomised controlled trial. Diabetologia. 2018 Jul;61(7):1548-1559. doi: 10.1007/s00125-018-4618-y. Epub 2018 Apr 26. PMID 29696296
- [Derived] Stomby A, Otten J, Ryberg M, Nyberg L, Olsson T, Boraxbekk CJ. A Paleolithic Diet with and without Combined Aerobic and Resistance Exercise Increases Functional Brain Responses and Hippocampal Volume in Subjects with Type 2 Diabetes. Front Aging Neurosci. 2017 Dec 4;9:391. doi: 10.3389/fnagi.2017.00391. eCollection 2017. PMID 29255413
- [Derived] Otten J, Stomby A, Waling M, Isaksson A, Tellstrom A, Lundin-Olsson L, Brage S, Ryberg M, Svensson M, Olsson T. Benefits of a Paleolithic diet with and without supervised exercise on fat mass, insulin sensitivity, and glycemic control: a randomized controlled trial in individuals with type 2 diabetes. Diabetes Metab Res Rev. 2017 Jan;33(1):10.1002/dmrr.2828. doi: 10.1002/dmrr.2828. Epub 2016 Jun 30. PMID 27235022